CLINICAL TRIAL: NCT00002630
Title: HIGH-DOSE MELPHALAN CHEMOTHERAPY AND TOTAL BODY RADIATION WITH PERIPHERAL BLOOD STEM-CELL RECONSTITUTION FOR PATIENTS WITH RELAPSING MULTIPLE MYELOMA
Brief Title: High-Dose Melphalan, Total-Body Irradiation, and Peripheral Stem Cell Transplantation in Treating Patients With Multiple Myeloma in First Relapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Morie Gertz, M.D., Mayo Clinic Cancer Center
Purpose: Treatment
Other Study IDs: CDR0000064030; P30CA015083 (NIH); 928003 (Other: Mayo Clinic Cancer Center); V95-0613 (Other: NCI CTRP)
Record Dates: First submitted 1999-11-01; First posted 2004-07-29 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Filgrastim; Cyclophosphamide; Melphalan; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Drug: cyclophosphamide
Drug: melphalan
Procedure: peripheral blood stem cell transplantation
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining peripheral stem cell transplantation with chemotherapy and radiation therapy may allow the doctor to give higher doses of radiation and chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of high-dose melphalan plus total-body irradiation and peripheral stem cell transplantation in treating patients with multiple myeloma in first relapse.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess bone marrow reconstitution and peripheral blood cell counts of patients with multiple myeloma treated with high-dose melphalan (L-PAM) and total-body irradiation (TBI) followed by peripheral blood stem cell (PBSC) rescue. II. Assess the efficacy of intravenous L-PAM and TBI for treatment of relapsing/refractory myeloma. III. Assess the tolerability and toxicity of this regimen in patients with relapsing multiple myeloma. IV. Assess response rate and survival of relapsing/refractory patients treated with this regimen.

OUTLINE: Prior to entry, patients will have received 3 monthly courses of standard VAD followed by PBSC collection on Regimen A; those who responded to VAD continue standard VAD to best response and upon relapse (on or off therapy) proceed to Regimen B. Patients with no response to 3 courses of VAD and those with no response to an alkylating-based regimen proceed immediately to Regimen B following PBSC collection. The following acronyms are used: CTX Cyclophosphamide, NSC-26271 G-CSF Granulocyte Colony Stimulating Factor (Amgen), NSC-614629 L-PAM Melphalan, NSC-8806 PBSC Peripheral Blood Stem Cells VAD Vincristine/Doxorubicin/Dexamethasone TBI Total Body Irradiation Regimen A: Stem Cell Mobilization/Harvest. CTX; G-CSF. Regimen B: Single-Agent Myeloablative Chemoradiotherapy with Stem Cell Rescue. L-PAM; TBI (Co60 or linear accelerators of 4 MV or greater); with PBSC.

PROJECTED ACCRUAL: If 9 or fewer or 20 or more responses are seen in the first 50 patients treated, the study will be discontinued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Multiple myeloma confirmed by bone marrow plasmacytosis and with measurable M-component in the serum or urine by immunoelectrophoresis or immunofixation No Stage I myeloma No smoldering multiple myeloma Refractory to or in first relapse following an initial response to VAD (vincristine/doxorubicin/dexamethasone), with relapse defined as any of the following: 50% increase above the lowest remission level of serum or urine M-protein while on therapy 25-50% increase above the lowest remission level of serum or urine M-protein associated with either: Hypercalcemia (greater than 11 mg/dl) Hb decrease of 2 g/dl attributable to increasing marrow plasmacytosis Appearance of new lytic lesions Calcium no greater than 11 mg/dl No myeloma meningitis No plasma cell leukemia

PATIENT CHARACTERISTICS: Age: 18 to 65 Performance status: ECOG 0-2 Hematopoietic: WBC greater than 500 (after G-CSF) Platelets greater than 25,000 Hepatic: Bilirubin no greater than 2.0 mg/dl Renal: Creatinine no greater than 2.0 mg/dl Cardiovascular: No NYHA class II-IV disease Pulmonary: DLCO at least 50% of predicted FVC at least 75% of predicted FEV1 at least 60% of predicted Other: No uncontrolled infection No active fungal infection No fever No prior malignancy within 5 years except: Basal cell skin cancer In situ carcinoma of the cervix No pregnant or nursing women

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior biological response modifiers allowed Chemotherapy: No time limit between cytotoxic therapy and protocol treatment Prior cumulative melphalan dose less than 300 mg Endocrine therapy: Corticosteroids for hypercalcemia allowed Radiotherapy: Prior radiotherapy allowed Prior pelvic radiotherapy allowed, but patients with such therapy are unlikely to have adequate PBSC harvested Surgery: Not specified

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 1993-06; Primary Completion 1999-02 (Actual); Study Completion 2001-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morie A. Gertz, MD, Study Chair — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mayo Clinic Cancer Center, Rochester, Minnesota

REFERENCES:
- [Background] Porrata LF, Gertz MA, Inwards DJ, Litzow MR, Lacy MQ, Tefferi A, Gastineau DA, Dispenzieri A, Ansell SM, Micallef IN, Geyer SM, Markovic SN. Early lymphocyte recovery predicts superior survival after autologous hematopoietic stem cell transplantation in multiple myeloma or non-Hodgkin lymphoma. Blood. 2001 Aug 1;98(3):579-85. doi: 10.1182/blood.v98.3.579. PMID 11468153
- [Background] Rajkumar SV, Fonseca R, Dispenzieri A, Lacy MQ, Witzig TE, Lust JA, Larson D, Therneau TM, Kyle RA, Litzow MR, Greipp PR, Gertz MA. Effect of complete response on outcome following autologous stem cell transplantation for myeloma. Bone Marrow Transplant. 2000 Nov;26(9):979-83. doi: 10.1038/sj.bmt.1702640. PMID 11100277
- [Result] Gertz MA, Lacy MQ, Inwards DJ, Gastineau DA, Tefferi A, Chen MG, Witzig TE, Greipp PR, Litzow MR. Delayed stem cell transplantation for the management of relapsed or refractory multiple myeloma. Bone Marrow Transplant. 2000 Jul;26(1):45-50. doi: 10.1038/sj.bmt.1702445. PMID 10918404
- [Result] Gertz MA, Lacy MQ, Inwards DJ, Chen MG, Pineda AA, Gastineau DA, Greipp PR, Lust JA, Tefferi A, Witzig TE, Kyle RA, Litzow MR. Early harvest and late transplantation as an effective therapeutic strategy in multiple myeloma. Bone Marrow Transplant. 1999 Feb;23(3):221-6. doi: 10.1038/sj.bmt.1701559. PMID 10084252
- [Result] Rajkumar S, Fonseca R, Lacy M, Witzig T, Lust J, Greipp P, Therneau T, Kyle R, Litzow M, Gertz M. Abnormal cytogenetics predict poor survival after high-dose therapy and autologous blood cell transplantation in multiple myeloma. Bone Marrow Transplant. 1999 Sep;24(5):497-503. doi: 10.1038/sj.bmt.1701943. PMID 10482933
- [Result] Rajkumar SV, Fonseca R, Dewald GW, Therneau TM, Lacy MQ, Kyle RA, Greipp PR, Gertz MA. Cytogenetic abnormalities correlate with the plasma cell labeling index and extent of bone marrow involvement in myeloma. Cancer Genet Cytogenet. 1999 Aug;113(1):73-7. doi: 10.1016/s0165-4608(99)00009-6. PMID 10459351
- [Result] Rajkumar SV, Fonseca R, Lacy MQ, Witzig TE, Lust JA, Greipp PR, Therneau TM, Kyle RA, Litzow MR, Gertz MA. Autologous stem cell transplantation for relapsed and primary refractory myeloma. Bone Marrow Transplant. 1999 Jun;23(12):1267-72. doi: 10.1038/sj.bmt.1701805. PMID 10414914
- [Result] Rajkumar SV, Fonseca R, Lacy MQ, Witzig TE, Lust JA, Greipp PR, Therneau TM, Kyle RA, Litzow MR, Gertz MA. Beta2-microglobulin and bone marrow plasma cell involvement predict complete responders among patients undergoing blood cell transplantation for myeloma. Bone Marrow Transplant. 1999 Jun;23(12):1261-6. doi: 10.1038/sj.bmt.1701787. PMID 10414913